CLINICAL TRIAL: NCT00890864
Title: Pilot Study of the Feasibility and Acceptability of Randomising the phasing-in of the Age Extension of the NHS Breast Screening Programme in England
Brief Title: Pilot Study: Age Extension of NHS Breast Screening Programme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: NHS Cancer Screening Programmes (Unknown); Department of Health, United Kingdom (Other Government)
Responsible Party: Heather House, Clinical Trials and Research Governance, Oxford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 09/H0710/2; ISRCTN50037017
Record Dates: First submitted 2009-01-26; First posted 2009-04-30 (Estimated); Last update posted 2010-07-19 (Estimated); Status verified 2010-07

CONDITIONS: Routine Mammography
Keywords: Breast screening; Mammogram; Routine screening programme

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Women aged 47-49 invited for breast screening
  Interventions: Other: Invitation for breast screening
- 2 (Active Comparator): Women aged 71-73 invited for breast screening
  Interventions: Other: Invitation for breast screening

INTERVENTIONS:
Other: Invitation for breast screening — Invitation for breast screening to women in different age groups
  Other Names: Invitation for mammogram

SUMMARY:
The purpose of this pilot study is to assess the feasibility and acceptability of randomising the phasing-in of the age extension of the NHS Breast Screening Programme in six volunteer sites in different areas of England.

DETAILED DESCRIPTION:
Currently all women are invited for breast screening between the ages of 50 and 70. In 2007 the Cancer Reform Strategy announced that from 2012 the NHS Breast Screening Programme would be extended to cover women between the ages of 47 and 73. This means that all women will get two extra screening invitations in their lifetime. It also means that all women will get their first invitation before age 50. As capacity does not allow for full immediate roll out across the whole of England, the age extension will be phased-in with full coverage from 2012. Randomising this phasing-in would provide unbiased evidence on the extent to which it is beneficial to extend the age range for breast screening and whether an extra screen at younger or older ages is more worthwhile. To date there is no clear evidence on this as no trial has looked at the added value of one extra screen within an existing screening programme. This pilot study will assess the feasibility and acceptability of randomising the phasing-in of the age extension in six volunteer sites in different areas of England.

ELIGIBILITY:
Inclusion Criteria:

* female, and living in one of the 6 pilot areas, and
* aged 47-49 or 71-73 years, and
* in a screening invitation batch that includes their age group.

Ages: 47 Years to 73 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36000 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Screening uptake among women invited for screening in the extended age groups | One year

SECONDARY OUTCOMES:
Workload associated with inviting these new age groups for screening | One year
Self-referrals among women in the pilot areas aged 47-49 or 71-73 but who were not invited for screening | One year

CONTACTS AND LOCATIONS:
Overall Officials: Julietta Patnick, BA (Hons), Principal Investigator — NHS Cancer Screening Programmes; also, Oxford University

REFERENCES:
- [Derived] Moser K, Sellars S, Wheaton M, Cooke J, Duncan A, Maxwell A, Michell M, Wilson M, Beral V, Peto R, Richards M, Patnick J. Extending the age range for breast screening in England: pilot study to assess the feasibility and acceptability of randomization. J Med Screen. 2011;18(2):96-102. doi: 10.1258/jms.2011.011065. PMID 21852703